CLINICAL TRIAL: NCT05640180
Title: Finerenone on Top of SGLT2is: A coMparatIve Hybrid Study Based oN RCT/RWE Data Of Patients With Chronic Kidney Disease Associated With Type 2 Diabetes
Brief Title: An Observational Study Called FLAMINgO to Learn More About the Treatment Combination of Finerenone and SGLT2 Inhibitors in People With Long-term Kidney Disease (Chronic Kidney Disease) Together With Type 2 Diabetes by Using Routine Medical Care Data and Past Clinical Study Results
Acronym: FLAMINGO
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22304
Record Dates: First submitted 2022-11-21; First posted 2022-12-07 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Chronic Kidney Disease; Type 2 Diabetes
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus, Type 2 | interventions — finerenone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- External control arm (ECA): ECA built from patients from Optum® Electronic Health Records (EHR) real world data (RWD) that closely match Sodium/glucose cotransporter-2 inhibitors (SGLT2i) subgroups from the randomized clinical trials (RCTs).
  Interventions: Drug: Sodium-glucose cotransporter-2 inhibitors (SGLT2i)
- Internal control arm (ICA): ICA built from participants from two RCTs called FIDELIO-DKD and FIGARO-DKD pooled for the FIDELITY analyses. FIDELIO-DKD/FIGARO-DKD placebo controls treated with SGLT2is at baseline.
  Interventions: Drug: Finerenone (Kerendia, BAY94-8862); Drug: Sodium-glucose cotransporter-2 inhibitors (SGLT2i)

INTERVENTIONS:
Drug: Finerenone (Kerendia, BAY94-8862) — Retrospective cohort analysis using randomized clinical trials data.
  Groups: Internal control arm (ICA)
Drug: Sodium-glucose cotransporter-2 inhibitors (SGLT2i) — Retrospective cohort analysis using United States Optum Electronic Health Records data.

SUMMARY:
This is an observational study, in which data from the past of people with chronic kidney disease (CKD) together with type 2 diabetes (T2D) are studied. The participants in this study were treated in the past with a type of drug called SGLT2 inhibitor alone or with SGLT2 inhibitors in combination with finerenone.

In observational studies, only observations are made without specified advice or interventions.

CKD is a long-term progressive decrease in the kidneys' ability to work properly. In people with T2D, the body does not make enough of a hormone called insulin, or does not use insulin well enough, resulting in high blood sugar levels that can cause damage to the kidneys. Chronic kidney disease often occurs together with / as a consequence of type 2 diabetes.

SGLT2 inhibitors lower blood sugar levels by increasing sugar removal from the blood into the urine. SGLT2 inhibitors are the standard of care (SOC) treatment for CKD and T2D. SOC is the treatment that medical experts consider most appropriate for a disease. The drug finerenone works by blocking certain proteins, called mineralocorticoid receptors.

By doing this, finerenone reduces damage to kidneys, heart and blood vessels. It is available and approved for doctors to prescribe to people with CKD together with T2D.

Results from two earlier clinical studies called FIDELIO-DKD and FIGARO-DKD in participants with CKD together with T2D are available. These results suggest that the treatment combination of finerenone and SGLT2 inhibitors may work better than taking SGLT2 inhibitors alone. The treatment combination may further slow down a worsening of the participants'

* kidney disease
* heart and blood circulation health.

Due to a limited number of participants treated with SGLT2 inhibitors alone however, the data from the two earlier studies does not allow to draw conclusions.

The main objective of this study is to combine additional real world data from SGLT2 inhibitor users with the study data from the earlier studies to get clearer results. Before combining the data however, statistical tests need to prove that this is allowed. If this is the case, the new combined "control" data can be compared with the data from the combination treatment group from the earlier studies. This will allow the researchers to get more proof and draw conclusions of how well the treatment combination works compared to SGLT2 inhibitors alone.

The real world data will come from a database called Optum. It will cover the period from January 2013 to September 2021. Only data from people who are similar to the participants of the control group of the earlier studies and meet certain criteria will be selected.

Only data from the past is collected and studied. There are no required visits or tests in this study.

ELIGIBILITY:
Inclusion Criteria:

* FIDELIO-DKD patients: Participants with a clinical diagnosis of DKD based on either of the following criteria at the Run-in and Screening Visit: Persistent high albuminuria or Persistent very high albuminuria.
* FIGARO-DKD patients: Participants with a clinical diagnosis of DKD based on either of the following criteria at the Run-in and Screening Visit: Persistent high albuminuria or Persistent very high albuminuria.
* Men or women aged 18 years and older
* Women of childbearing potential can only be included in the study if a pregnancy test is negative at the Screening Visit and if they agree to use adequate contraception.
* Diagnosed with type 2 diabetes.
* Prior treatment with Angiotensin-converting-enzyme inhibitors (ACEIs) and Angiotensin receptor blockers (ARBs) as follows:

  * For at least 4 weeks prior to the Run-in Visit, subjects should be treated with either an ACEI or ARB, or both
  * Starting with the Run-in Visit, subjects should be treated with only an ACEI or ARB
  * For at least 4 weeks prior to the Screening Visit, subjects should be treated with the maximum tolerated labeled dose (but not below the minimal labeled dose) of only an ACEI or an ARB (not both) preferably without any adjustments to dose or choice of agent or to any other antihypertensive or antiglycemic treatment.
* Serum potassium ≤4.8 mmol/L at both the Run-in and the Screening Visit.
* SGLT2 inhibitor use at baseline: Canagliflozin, Dapagliflozin, Empagliflozin, Ertugliflozin, Ipragliflozin, Luseogliflozin, Tofogliflozin.

Exclusion Criteria:

* Known significant non-diabetic renal disease, including clinically relevant renal artery stenosis.
* Urine Albumin-Creatinine Ratio (UACR) >5000 mg/g (>565 mg/mmol) at the Run-in Visit or Screening Visit.
* Hemoglobin A1C (HbA1c) > 12% (> 108 mmol/mol) at the Run-in Visit or Screening Visit.
* Uncontrolled arterial hypertension with mean sitting systolic blood pressure (SBP) ≥170 mmHg or mean sitting diastolic blood pressure (DBP) ≥110 mmHg at the Run-in Visit or mean sitting SBP ≥160 mmHg or mean sitting DBP ≥100 mmHg at the Screening Visit.
* Mean SBP < 90 mmHg at the Run-in Visit or at the Screening Visit.
* Subjects with a clinical diagnosis of chronic heart failure with reduced ejection fraction (HFrEF) and persistent symptoms (New York Heart Association class II - IV) at the Run-in Visit (class 1A recommendation for MRAs).
* Stroke, transient ischemic cerebral attack, acute coronary syndrome, or hospitalization for worsening heart failure, in the last 30 days prior to the Screening Visit.
* Dialysis for acute renal failure within 12 weeks prior to the Run-in Visit.
* Renal allograft in place or a scheduled kidney transplant within the next 12 months from the Run-in Visit.
* Addison's disease.
* Hepatic insufficiency classified as Child-Pugh C.
* Concomitant therapy with eplerenone, spironolactone, any renin inhibitor, or potassium-sparing diuretic which cannot be discontinued at least 4 weeks prior to the Screening Visit.
* Concomitant therapy with both ACEI and ARBs which cannot be discontinued for the purpose of the study.
* Concomitant therapy with potent cytochrome P450 isoenzyme 3A4 (CYP3A4) inhibitors or inducers (to be stopped at least 7 days before randomization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The randomized clinical trials (RCT) source population is comprised from participants who were enrolled in the FIDELIO-DKD and FIGARO-DKD trials, pooled for the FIDELITY analyses. The source population for the real world (RW) cohort are patients in the Optum® Electronic health record (EHR) database, which includes longitudinal patient-level medical record data for ~97 million patients across the United States dating back to January 1st, 2007.
Sampling Method: Non-Probability Sample
Enrollment: 17847 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Time to the first occurrence of the composite endpoint of onset of kidney failure, a sustained decrease of eGFR ≥ 40% from baseline over at least 4 weeks, or renal death | From randomization up until the first occurrence of the primary renal composite endpoint, or censoring at the end of the study, with a maximum follow-up time of 48 months
Time to first occurrence of the composite endpoint of Cardiovascular (CV) death or non-fatal CV event (i.e. myocardial infarction, stroke, or hospitalization for heart failure) | From randomization up until the first occurrence of the key secondary CV composite endpoint, or censoring at the end of the study, with a maximum follow-up time of 48 months

SECONDARY OUTCOMES:
Time to all-cause hospitalization | From randomization up until the first occurrence of the hospitalization due to any cause, or censoring at the end of study, with a maximum follow-up time of 48 months
Time to all-cause mortality | From randomization up until death due to any cause, or censoring at the end of the study, with a maximum follow-up time of 48 months
Change in urine albumin-creatinine ratio (UACR) from baseline to Month 4 | From baseline to Month 4
Time to first occurrence of the following composite endpoint: onset of kidney failure, a sustained decrease in eGFR of ≥ 57% from baseline over at least 4 weeks or renal death | From randomization up until the first occurrence of the composite primary endpoint, or censoring at the end of the study, with a maximum follow-up time of 48 months

CONTACTS AND LOCATIONS:
Locations (1):
- Bayer, Whippany, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.